CLINICAL TRIAL: NCT06733337
Title: Special Investigation of TALZENNA Capsules - Study on BRCA Mutation-Positive Metastatic Castration-Resistant Prostate Cancer -
Brief Title: A Study to Learn About the Safety of TALZENNA in People With Prostate Cancer.
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3441050
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: BRCA mutation-positive; metastatic castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to learn about the safety of TALZENNA in patients with BRCA mutation-positive metastatic castration-resistant prostate cancer. BRCA mutation positive means any changes to the BRCA gene. Metastasis means the cancer that has spread to other parts of the body. Castration-resistant prostate cancer means the prostate cancer that keeps growing even when the amount of male sex hormone in the body is reduced to very low levels. Prostate is a male sex organ.

The study is seeking for participants:

* with BRCA mutation-positive metastatic castration-resistant prostate cancer
* who have not used this study medicine before. All patients in this study will receive TALZENNA according to the prescriptions.

Patients will be followed up to 52 weeks (12 months) from the day of start of treatment start (Day 1). However, in cases where treatment has been completed or stopped less than 52 weeks (12 months) after the start of giving study medicine, the participants will be checked until completion (discontinuation) of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BRCA mutation-positive metastatic castration-resistant prostate cancer
* No history of previous use of this drug

Exclusion Criteria:

* None

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The target disease, prostate cancer, is specific to male.
Study Population: Patients who satisfy the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-07-11 (Actual); Primary Completion 2029-06-22 (Estimated); Study Completion 2029-06-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions | Up to 52 weeks
  For adverse drug reactions corresponding to myelosuppression, interstitial lung disease, thromboembolism, and secondary malignant tumour, the incidence, time of onset, grade, outcome etc. will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Japan, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441050